CLINICAL TRIAL: NCT02728349
Title: Phase 1 Trial of Tolerance and Pharmacokinetic of Chlorogenic Acid for Injection in the Advanced Glioblastoma Patients
Brief Title: Tolerance and Pharmacokinetic Study of Chlorogenic Acid to Advanced Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan J.Z. Bio-chemical Science and Technology Development Co., Ltd (Industry)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYS-I-03
Record Dates: First submitted 2016-03-28; First posted 2016-04-05 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2017-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Chlorogenic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chlorgenic acid, Treatment, powder (Experimental): Chlorogenic acid for injection(30mg/bottle) is white or off-white freeze-dried lump or powder,it can be easily dissolved in water, which solubility is 20%.
  Interventions: Drug: Chlorogenic acid

INTERVENTIONS:
Drug: Chlorogenic acid — Chlorogenic acid for injection is polyphenols, micromolecular and un-endogenous substance. It might play the role of cancer treatment via balancing tumor micro-environmental immune status according to the stability and rationality of immunodeficiency and endogenous immune material expression around the tumor. Chlorogenic acid for injection is made from chlorogenic acid (purity≥98%) which is extracted from folium cortex eucommiae.Chlorogenic acid and its preparations have not been reported as chemical drug and marketed around the world.

SUMMARY:
The purpose of this study:

Determining the Maximum Tolerated Dose (MTD), Dose-Limiting Toxicity (DLT), pharmacokinetics characteristic, and dosage regimen of phase II/III of Chlorogenic acid for injection in the advanced Glioblastoma Patients ;

DETAILED DESCRIPTION:
1. Investigate the tolerance of Chlorogenic acid for injection in human body, determine the Maximum Tolerated Dose (MTD) and Dose-Limiting Toxicity (DLT) of Chlorogenic acid for injection in the advanced Glioblastoma Patients ;
2. Determine the human pharmacokinetics characteristic of Chlorogenic acid for injection;
3. Preliminary observation the effectiveness and effective dose;
4. Provide the basis for the dosage regimen of phase II/III.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologic or/and FNAC confirmation of advanced glioblastoma(WHO,III-IV grade) but without effective treatment or with treatment failure;
2. Between 18 and 65 years of age, KPS≥40;
3. According to RANO(2010), the parents will be eligible if one of the following conditions apply: steroid dose increased or stable,the enhanced tumor lesion increased more than 25%; the unenhanced tumor lesion increased because of the progressive tumor,even if the lesion was unmeasurable.
4. Life expectancy of at least three (3) months at the enrollment;
5. Patients who have sufficient baseline organ function and whose laboratory data can meet the following criteria at the enrollment:

1)PLT count≥100×10~9/L, 2)WLB count≥4.0×10~9/L and ≤12×10~9/L, 3)Neutrophil granulocyte count≥2.0×10~9/L, 4)HGB count≥90g/L, 5)Total bilirubin <=1.5 times of ULN, 6)ALT/AST ≤2.5 times of ULN, 7)SCr≤1.5 times of ULN, 8)Normal ECG with LVEF (≥50%) measured by echocardiography; 6.Female patients with negative pregnant test, and male/female patients of reproductive age without pregnancy planning in the next 12 months; 7.Volunteered for the phase 1 trial and sign the informed consent without protest;

Exclusion Criteria:

1. Patients who have received large area radiotherapy （>30% marrow capacity）;
2. Without pathologic or/and FNAC confirmation of advanced glioblastoma;
3. Patients who has primary immunodeficiency diseases；
4. Patients who suffer from other serious complication, such as uncontrollable infection, myocardial infarction within the past 6 months at the enrollment , uncontrollable hypertension ,thromboembolism and etc.;
5. Patients who have received the therapy of chemotherapy or radical radiotherapy within 4 weeks before enrollment;
6. Patients who have used nitrosoureas drug or mitomycin within 6 weeks or tyrosine kinase inhibitor within 2 weeks before enrollment;
7. Patients who have received therapy of major surgery within 4 weeks or biopsy surgery within 2 weeks before enrollment;
8. Patients who experience grade 2 or more than grade 2 toxicity caused by the past therapies;
9. Patients who have history of drug abuse;
10. Uncontrollable psychopaths；
11. Uncontrollable diabetes；
12. Pregnant or breast-feeding women, or patients(male and female) who have pregnancy plan;
13. Patients who had received a therapy of another investigational drug within 12 weeks or patients who are still in another clinical trial at the enrollment;
14. Known active hepatitis B/hepatitis C, positive HIV/ syphilis antibody;
15. Patient who need long term treatment of cortical hormone or other immunosuppressive drugs such as visceral organ transplanters;
16. Allergic to the investigational drug;
17. Other patients judged ineligible for enrollment in the study by the investigator (sub-investigator).
18. Patients who have received the therapy of adrenal steroid hormones within 1 week before enrollment or will receive the therapy for a long period time，except for Corticosteroid nasal spray，Inhaled Steroid and Topical steroids .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Within the first 30 days after the first dose of chlorogenic acid
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0，grade ≥3 (DLT) | Within the first 30 days after the first dose of chlorogenic acid
Maximum Tolerated Dose | Within the first 30 days after the first dose of chlorogenic acid
Area under the plasma concentration versus time curve (AUC) of chlorogenic acid | Within the first 30 days after the first dose of chlorogenic acid
Peak Plasma Concentration (Cmax) of chlorogenic acid | Within the first 30 days after the first dose of chlorogenic acid

SECONDARY OUTCOMES:
Improvement in cancer-related symptoms | Within 1 year after the first dose of chlorogenic acid
disease control rate(DCR) | Within the first 30 days after the first dose of chlorogenic acid
objective response rate (ORR) | Within the first 30 days after the first dose of chlorogenic acid
progress free survival(PFS) | Within the first 30 days after the first dose of chlorogenic acid
overall survival (OS) | Within the first 30 days after the first dose of chlorogenic acid
Improvement in quality of life | Within 1 year after the first dose of chlorogenic acid

OTHER OUTCOMES:
Changing in number of red blood cell | Within 1 year after the first dose of chlorogenic acid
Changing in cytokines in peripheral blood | Within 1 year after the first dose of chlorogenic acid
Changing in level of hemoglobin | Within 1 year after the first dose of chlorogenic acid
Changing in lymphocyte subsets | Within 1 year after the first dose of chlorogenic acid

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital,Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No